CLINICAL TRIAL: NCT02284776
Title: Preliminary Evaluation Study of Therapeutic Education on Overweight People in Addition to a Hydrotherapeutic Cure at the Thermal Baths of Brides-les-Bains
Brief Title: Preliminary Evaluation Study of Therapeutic Education on Overweight People in Addition to a Hydrotherapeutic Cure
Acronym: Educatherm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Pasteur de Lille (Other)
Collaborators: Association Francaise pour la Recherche Thermale (Other); Société des Etablissements Thermaux de Brides-les-Bains et Salins-les-Bains (Unknown); Centre d'Investigation Clinique 9301 INSERM-CHRU de Lille (Unknown)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, medical doctor specializing in endocrinology and metabolic diseases, Institut Pasteur de Lille
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2013-A00226-43
Record Dates: First submitted 2013-10-30; First posted 2014-11-06 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Obesity
Keywords: Therapeutic education
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Témoin (No Intervention): No treatment.
- Action (Experimental): People in hydrotherapeutic cure are following a program of Therapeutic Education. This program includes dietary advice, physical activities, behavior advice in order to change the lifestyle of the obese people.
  Interventions: Behavioral: Therapeutic education

INTERVENTIONS:
Behavioral: Therapeutic education — People in hydrotherapeutic cure are following a program of Therapeutic Education. This program includes dietary advice, physical activities, behavior advice in order to change the lifestyle of the obese people.
  Arms: Action

SUMMARY:
The goal of this study is to assess the effect of a therapeutic education program in addition of a hydrotherapeutic cure on obese patients.

The therapeutic education program at the thermal baths of Brides-les-Bains is composed of a dietary follow-up, a physical activities program, working group.

DETAILED DESCRIPTION:
The participants are people that come to the thermal baths in order to follow an hydrotherapeutic cure (of about 3 weeks). For the Action group, they also follow a course of therapeutic education where they are given advices on how they should eat and have a regular physical activity.

This therapeutic education in addition of the hydrotherapeutic cure should help them lose weight and not gain in again.

The participants are followed for 18 months (17 months after leaving the thermal baths).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) over 27 kg/m² (or equal)
* Has a valid email address, has access to the internet and to a telephone line
* Has a domestic scale compatible with its weight
* Signed the consent form
* Susceptible to accept the obligations generated by the study
* Has a health insurance

Exclusion Criteria:

* Has a progressive illness at the time of the study (cancer, neurodegenerative disease...)
* Is pregnant
* Follows the hydro-therapeutic cure in order to cure rheumatism
* Trying to lose weight prior to a surgery
* Has a diagnosed eating disorder
* Has no physical activity due to a handicap or a serious osteoarthritis
* Has taken a weight-loss drug (Orlistat) in the past month or will likely do so in the future
* Is taking a Desmopressin-based drug
* Is unable to understand or follow the protocol
* Is deprived of liberty
* Is under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-02 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Change in the weight between the end of the hydrotherapeutic cure and 5 months after the hydrotherapeutic cure | People's weight in between the end of hydrotherapeutic cure and 5 months after hydrotherapeutic cure
  People weight themselves on a domestic scale.

SECONDARY OUTCOMES:
Evolution of the weight. | 0 ; 3 weeks ; 6 months ; 12 months ; 18 months
  People weight themselves on a domestic scale.
Quality of life | 0 ; 3 weeks ; 6 months ; 12 months
  Assessed with the Short SF-36 questionnaire.
Physical activity | 0 ; 3 weeks ; 6 months ; 12 months
  Assessed with the Ricci-Gagnon questionnaire.
Individual's readiness to change | 0 ; 3 weeks ; 6 months ; 12 months
  Assessed with the Prochaska questionnaire.
Visual and analogical scale for general and psychological well-being and body discomfort. | 0 ; 3 weeks ; 6 months ; 12 months
  Participants mark down on a 10cm scale how they feel.
Felling about the body | 0 ; 3 weeks ; 6 months ; 12 months
  Questionnaire on how the participants feel about their body.
Dietary habits | 0 ; 3 weeks ; 6 months ; 12 months
  Questionnaire about the dietary habits of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Lecerf, MD, Principal Investigator — Institut Pasteur de Lille
Locations (1):
- SET Brides-les-Bains, Brides-les-Bains, Savoir, France